CLINICAL TRIAL: NCT06840587
Title: Transitional Care for Skilled Nursing Facility Patients With Alzheimer's Disease and Related Dementias and Their Caregivers: a Cluster Randomized Trial
Brief Title: Connect-Home: Alzheimer's Disease and Related Dementias
Acronym: CH-ADRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-2766; 2R01NR017636-05A1 (NIH)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Before enrollment of SNF patients and caregivers, randomization of the 12 SNFs will be conducted by blinded study staff who will use codes to conceal allocation and randomly assign SNFs in a 1:1 ratio to intervention and control arms. Study staff masked to study arm will assess outcomes, in a telephone-based interview with caregivers in both arms, 30 days after SNF discharge, this is for research purposes only. Research coordinators (RCs) will conduct 30-day electronic health record (EHR) reviews after dyads complete study participation, as EHR content has the potential to reveal study arm assignment. As with most behavioral clinical interventions, participants and care providers cannot be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connect-Home ADRD Intervention (Experimental): The Connect-Home ADRD Intervention will include:
  1. Support for SNF staff delivery of transitional care processes including a ADRD transition plan and booklet, caregiver training and engagement, and handoff of care to community providers and Dementia Caregiving Specialist.
  2. Support for patients and caregivers provided by the Dementia Caregiving Specialist in three follow-up supportive telephone calls within 30 days of SNF discharge.
  Interventions: Behavioral: Connect-Home ADRD
- Standard Care - Control Group (No Intervention): Patient and caregiver dyad randomized to the control arm will receive usual SNF and post-discharge care.

INTERVENTIONS:
Behavioral: Connect-Home ADRD — Connect-Home ADRD will introduce new structure and processes to support SNF staff delivery of transitional care for transitions to home, assisted living, or long-term care, and post-discharge transitional care by the Dementia Caregiving Specialist.
  Arms: Connect-Home ADRD Intervention

SUMMARY:
This study is a parallel arm, cluster randomized trial (CRT) to test the efficacy of Connect-Home ADRD, a transitional care intervention focusing on Skilled Nursing Facility (SNF) patients with Alzheimer's disease and dementias and their caregivers during transitions from SNFs to home, assisted, living, and long-term care. The primary hypothesis is that the intervention will reduce caregiver strain (Aim 1) and patient neuropsychiatric symptoms (Aim 2).

DETAILED DESCRIPTION:
Connect-Home ADRD is a Donabedian-guided intervention that introduces new structure and processes to support Skilled Nursing Facility (SNF) staff delivery of transitional care for transitions to home, assisted living, or long-term care, and post-discharge transitional care by the Dementia Caregiving Specialist (DCS).

The research objective is to test the efficacy of Connect-Home ADRD, a transitional care intervention, targeting Skilled Nursing Facility (SNF) patients with Alzheimer's disease and related dementias (ADRD) and their primary caregivers who discharge home and other settings of care. The study will be set in 12 North Carolina SNFs and in the patient's discharge destination (during intervention periods only). Using a cluster-randomized trial design, twelve SNFs will be randomly allocated to an intervention group (N=6 SNFs) and to a control group (N=6 SNFs) by a study statistician masked to SNF identity. 360 dyads of SNF patients with ADRD and caregivers will be enrolled in 12 SNFs.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Ability to speak English
* Goal of discharge to home, assisted living, or long-term care
* Diagnosis of dementia
* Having a caregiver willing to participate

Caregivers:

* Ability to speak English
* Legally authorized representative (LAR) who also provides support for the person with ADRD

Inclusion criteria for SNFs:

* Location within 120 miles of UNC-Chapel Hill
* Admission of at least 75 SNF patients per year

Exclusion Criteria:

Patients:

* Planned hospital readmission for procedures or treatments within 30 days post enrollment.

Caregivers:

* LAR is a court-appointed guardian.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Caregiver Strain | 30 days after discharge from SNF
  Modified Caregiver Strain Index Score (MCSI): 13 yes-no items, measure indicators of caregiver strain over the past 30 days. Summary score ranges from 0-26, higher scores indicating greater strain.
Patient Neuropsychiatric Symptoms | 30 days after discharge from SNF
  Neuropsychiatric Inventory-Q (NPI-Q): 12 items on a 3-point scale, measures presence and severity of neuropsychiatric symptoms over the past 30 days. Summary score ranges from 0-36, higher scores associated with more severe symptoms.

SECONDARY OUTCOMES:
Caregiver Depression | 30 days after discharge from SNF
  Patient Health Questionnaire-8 (PHQ-8): 9 items on a 4-point scale, measures depressive symptoms over the past 30 days. Scores range from 0-27, higher scores indicate more depressive symptoms.
Preparedness for care transitions | 30 days after discharge from SNF
  Care Transitions Measure-15 (CTM-15): 15 items on a 4-point scale, measures self-reported knowledge to continue care after discharge. Summary score ranges from 0-100, higher scores associated with less acute care use after discharge.
Patient Quality of Life | 30 days after discharge from SNF
  Quality of Life in Alzheimer's Disease (QoL-AD): 13 items on a 4-point scale measuring caregiver-reported quality of life in people with ADRD over the past 30 days. Summary scores range from 13-52, with higher scores indicating higher quality of life.
Acute Care Use | 30 days after discharge from SNF
  Caregiver-reported days of emergency department and hospital use in 30 days after SNF discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Toles, PhD, RN, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 9 to 36 months following publication
Access Criteria: Data may be requested to achieve aims in an approved proposal if an investigator has approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.